CLINICAL TRIAL: NCT05008835
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of ACP-044 in Subjects With Pain Associated With Osteoarthritis of the Knee
Brief Title: Evaluate the Efficacy and Safety of ACP-044 in Subjects With Pain Associated With Osteoarthritis of the Knee
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated for business reasons.
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-044-005
Record Dates: First submitted 2021-08-10; First posted 2021-08-17 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Drug - ACP-044 Dose A (Experimental): ACP-044 Dose A
  Interventions: Drug: ACP-044 Dose A
- Drug - ACP-044 Dose B (Experimental): ACP-044 Dose B
  Interventions: Drug: ACP-044 Dose B
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACP-044 Dose A — Oral dose of ACP-044 Dose A
  Arms: Drug - ACP-044 Dose A
Drug: ACP-044 Dose B — Oral dose of ACP-044 Dose B
  Arms: Drug - ACP-044 Dose B
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of ACP-044 compared with placebo in the treatment of pain associated with osteoarthritis of the knee

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥18 and <65 years of age at the time of Screening
* Has a body mass index (BMI) ≤39 kg/m2 at Screening
* Confirmed history of pain associated with OA in the index knee
* Willing to maintain current activity and exercise levels throughout the study
* Willing and able to comply with clinic visits and study-related procedures
* Consent to allow all radiographs and medical/surgical/hospitalization records of care received elsewhere to be shared with the Investigator and third parties who will examine the images (i.e., central x-ray reader)

Exclusion Criteria:

* Pain anywhere else in the body which is greater than or equal to OA pain in the index knee, or likely to interfere with subject's assessment of pain throughout the study, as judged by the Investigator
* History or presence on imaging of knee arthropathy (osteonecrosis, subchondral insufficiency fracture, rapidly progressive OA type 1 or type 2), recent fall, injury, or trauma affecting the index knee, ligament tear, neuropathic joint arthropathy, knee dislocation (patella dislocation is eligible), extensive subchondral cysts, Baker's cyst, evidence of bone fragmentation or collapse, or primary metastatic tumor with the exception of chondromas, or pathological fractures during the Screening Period
* History or presence at Screening of non-OA inflammatory joint disease (e.g., rheumatoid arthritis, lupus erythematosus, psoriatic arthritis, pseudo-gout, gout, spondyloarthropathy, joint infections within the past 5 years, Paget's disease of the spine, pelvis, or femur, neuropathic disorders, multiple sclerosis, fibromyalgia, tumors or infections of the spinal cord, or renal osteodystrophy) or any condition that would interfere with the rating of OA pain
* Recent arthroscopic surgery within 1 month of Screening; or has any planned surgery or procedure during the study
* Use of monoamine reuptake inhibitors, tricyclic antidepressants, anticonvulsants, and/or serotonin norepinephrine reuptake inhibitors within 4 weeks prior to Screening
* Unwilling to discontinue current use of analgesic medication following Screening and to adhere to study requirements for rescue treatments (study-provided acetaminophen to be taken as needed with a maximum daily dose of 2500 mg), including, but not limited to, nonsteroidal anti-inflammatory drugs (NSAIDs), opioids, selective cyclooxygenase 2 inhibitors, acetaminophen, or combinations thereof, within 7 days or five half-lives of the drug prior to the Baseline Pain Assessment Period, whichever is longer
* Use of immediate- or extended-release or controlled-release opioids (e.g., oxycontin), transdermal fentanyl, or methadone within 3 months prior to Screening
* Use of opioids, for the treatment of pain other than OA of the knee, with a morphine equivalent dose of ≥30 mg per day for more than 2 days per week within 1 month prior to Screening
* Use of systemic (i.e., oral) corticosteroids or intra-articular corticosteroids in any joint within 30 days prior to the screening visit (topical, intranasal, and inhaled corticosteroids are permitted)
* Intra-articular injection of any approved (i.e., hyaluronic acid and corticosteroids) or unapproved treatments (e.g., platelet-rich plasma, capsaicin) into the index knee within 3 months of Screening
* Physical/occupational/chiropractic therapy for the lower extremities or acupuncture for the lower extremities within 30 days of Screening, or the need for such therapy during the study
* Has current evidence, or history within the previous 12 weeks prior to Screening, of a serious and/or unstable psychiatric, neurologic, cardiovascular, respiratory, gastrointestinal, renal, hepatic, hematologic, endocrinologic, or other medical disorder, that in the judgment of the Investigator and/or Medical Monitor would jeopardize the safe participation of the subject in the study
* Had a malignancy in the last year, with the exception of nonmetastatic basal cell of the skin or localized carcinoma in situ of the cervix

Additional inclusion/exclusion criteria apply. Patients will be evaluated at screening to ensure that all criteria for study participation are met. Patients may be excluded from the study based on these assessments (and specifically, if it is determined that their baseline health and psychiatric condition do not meet all pre-specified entry criteria).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-11-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Clinical Research Investment, LLC, Birmingham, Alabama
  - AOC-Research, Birmingham, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - BioSolutions Clinical Research Center, La Mesa, California
  - Velocity Clinical Research, North Hollywood, North Hollywood, California
  - Artemis Headlands, LLC, San Diego, California
  - TriWest Research Associates, LLC, San Diego, California
  - Encompass Clinical Research, Spring Valley, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - M&M Medical Center, Miami, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Orlando, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Precision Clinical Research,LLC, Sunrise, Florida
  - Conquest Research, Winter Park, Florida
  - Drug Studies America, Marietta, Georgia
  - Health Research Network II, LLC, Flossmoor, Illinois
  - Affinity Health Corp., Oak Brook, Illinois
  - Medisphere Medical Research Center, LLC, Evansville, Indiana
  - Velocity Clinical Research-Boise, Meridian Hills, Indiana
  - AMR Wichita West, Wichita, Kansas
  - Alliance for Multispecialty Research, LLC., Lexington, Kentucky
  - Bay State Clinical Trials, Watertown, Massachusetts
  - Healthcare Research Network, Inc., Hazelwood, Missouri
  - AMR Las Vegas, Las Vegas, Nevada
  - Drug Trials America, Inc., Hartsdale, New York
  - Upstate Clinical Research Associates, LLC, Williamsville, New York
  - Hightop Medical Research Center, Cincinnati, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Future Search Trials, Austin, Texas
  - Clinical Investigations of Texas,LLC, Plano, Texas
  - Spectrum Medical, Inc., Danville, Virginia
  - Health Research of Hampton Roads, Newport News, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening period of up to 4 weeks, patients were assessed for eligibility. Prohibited medication was to be discontinued. Eligible patients had to complete a Baseline Pain Assessment Period of about 7 days before randomization (allowed time window +3 days) to be instructed in the use of an electronic diary and to record pain scores and rescue medication use. Compliance with data recording was assessed for continued eligibility. Upon completion of this period, patients were randomised.
Groups:
- Placebo: Administration of ACP-044 matching placebo 4 times daily (morning, noon, evening, night)
- ACP-044 400 mg QID: Administration 4 times daily (morning, noon, evening, night) of 400 mg ACP-044 At each the morning and evening administration, patients received one placebo tablet and one tablet containing ACP-044 400 mg. At each the noon and night administration, patients received one tablet containing ACP-044 400 mg.
- ACP-044 800 mg BID: Administration 2 times daily (morning, noon, evening, night) of 800 mg ACP-044 At each the morning and evening administration, patients received 2 tablets containing ACP-044 400 mg. At each the noon and night administration, patients received one placebo tablet.
Period: Overall Study
Arm/Group | Placebo | ACP-044 400 mg QID | ACP-044 800 mg BID
Started | 21 | 20 | 20
Completed | 13 | 16 | 16
Not Completed | 8 | 4 | 4
Not completed — Adverse Event | 5 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 1
Not completed — Not further specified | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Population: All randomised patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ACP-044 400 mg QID | ACP-044 800 mg BID | Total
Number analyzed (Participants) | 21 | 20 | 20 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (5.02) | 58.1 (4.82) | 56.8 (5.31) | 57.2 (5.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 13 | 41
  Male | 7 | 6 | 7 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 5 | 14
  White | 14 | 17 | 14 | 45
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 20 | 61

OUTCOME MEASURES:

1. Primary Outcome: Weekly Average of the Daily Average Numeric Rating Scale (NRS) Pain Intensity Scores
Description: The 0-10 NRS consists of a single 11-point numeric scale, with 0 indicating no pain at all and 10 reflecting the worst pain imaginable.
  Due to the business decision to discontinue clinical development of ACP-044, this study was prematurely terminated. Efficacy was not evaluated in this study by using (planned) inferential statistics. For the purpose of results posting, changes in NRS over time are displayed using descriptive statistics.
Time Frame: 4 weeks
Population: All patients randomised and treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | ACP-044 400 mg QID | ACP-044 800 mg BID
Number analyzed (Participants) | 21 | 20 | 20
score on a scale
  Baseline: number analyzed (Participants) | 20 | 20 | 20
  Baseline | 5.4 (1.81) | 6.1 (1.12) | 5.6 (1.64)
  Week 1: number analyzed (Participants) | 15 | 17 | 16
  Week 1 | 3.1 (1.81) | 4.4 (2.24) | 4.6 (1.63)
  Week 2: number analyzed (Participants) | 12 | 15 | 17
  Week 2 | 3.0 (1.28) | 3.9 (2.26) | 4.2 (2.19)
  Week 3: number analyzed (Participants) | 10 | 11 | 12
  Week 3 | 2.9 (0.88) | 3.8 (2.36) | 4.2 (2.33)
  Week 4: number analyzed (Participants) | 0 | 2 | 1
  Week 4 |  | 4.0 (1.41) | 3.0 (NA) — Standard deviation not applicable if only a single patient is included in the assessment.

ADVERSE EVENTS:
Time Frame: AEs were planned to be reported from signing informed consent to the end of the follow-up period. Since the study was prematurely terminated, the AE reporting period was abbreviated and thus, AEs were assessed from signing the informed consent to the end of treatment, the mean (SD) duration of this period was 24.1 (8.2) days.
Arm/Group | Placebo | ACP-044 400 mg QID | ACP-044 800 mg BID
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 4/20 | 4/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=21) | ACP-044 400 mg QID (N=20) | ACP-044 800 mg BID (N=20)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the business decision to discontinue clinical development of ACP-044, this study was prematurely terminated. Instead of a planned number of 240 patients, only 61 patients were randomised. Due to these facts, efficacy was not evaluated in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to their own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the Sponsor for review and comment. The sponsor has 60 days to review and comment.

DOCUMENTS (2):
  • Study Protocol (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/35/NCT05008835/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT05008835/SAP_001.pdf